CLINICAL TRIAL: NCT03972865
Title: Cardiovascular Consequences and Risk of Ventricular Rhythm Disorder in Intense and Extended Physical Exercise
Brief Title: Cardiovascular Consequences in Intense and Extended Physical Exercise
Acronym: PHILIPPIDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL17_0385; 2018-A00237-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2022-01

CONDITIONS: Ventricular Arrythmia; Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants of the race (Experimental): Participants of the race are healthy triathlete volunteers who will participate in August 2019 in the Embrun (EmbrunMan) long-distance triathlon (Ironman)
  Interventions: Other: EmbrunMan race

INTERVENTIONS:
Other: EmbrunMan race — The EmbrunMan is a long-duration triathlon including 3.8 km of swimming, 188 km of cycling and 42.2 km of running, with a cumulative vertical drop of 4000 metres. Duration of the race varies between 10 hours and 16hours depending on the athletes' performance.

SUMMARY:
This research study because you participate in long distance triathlon of Embrun. In recent years, there has been a craze for races at increasingly longer distances (ultra-endurance) with risks to the cardiovascular system poorly identified. In the short term, cardiac functional ultrasonographic changes and disturbances of biomarkers such as troponin are reported in participants in long-term endurance trials, assuming myocardial remodeling and transient tissue damage leading to suffering or "heart fatigue". These constraints could, to the extreme, favor the development of arrhythmia at the atrial and ventricular stages. Cardiac alterations are nevertheless poorly characterized and the consequences, in particular the risk of ventricular rhythm disturbance, have not been studied.The aim of this study is to investigate the relationship between right ventricular functional abnormalities and the occurrence of ventricular rhythm disturbance, following intense and prolonged exercise, in healthy triathletes subjects.

DETAILED DESCRIPTION:
Background and rationale:

While regular and moderate physical activity is strongly recommended in reducing cardiovascular risk, the scientific community questions the potentially harmful effects of prolonged and intense physical activity. In the short term, functional ultrasonographic changes (systolic and diastolic) and disturbances of biomarkers such as troponin are reported in participants in long-term endurance trials, assuming myocardial remodeling and transient tissue damage leading to suffering or "heart fatigue". These constraints could, to the extreme, favor the development of arrhythmogenic foci at the atrial and ventricular stages, and at least, be responsible for a sudden death of the athlete. Adaptations of the athlete's heart have mainly been studied in the left ventricle but more and more studies are studying the right ventricle (RV). These alterations are nevertheless poorly characterized and the consequences including the risk of ventricular rhythm disorder have not been studied.

Primary and Secondary Objectives:

The primary objective is to test the existence of a relationship between RV functional abnormalities induced by intense and prolonged exercise, and the occurrence of ventricular ectopic beats (VEB) from RV. The secondary objectives are to characterize the respiratory impairment of this type of course and to study its relation with the functional anomalies of the RV and the occurrence of VEB.

Methodology:

This is a prospective study including male triathletes participating in the long-distance triathlon of Embrun in August 2019 (3.8 km of swimming, 188 km of cycling and 42.2 km of running), aged between 20 to 54 years years old. The criteria for non-inclusion are subjects with a history of heart disease or rhythm disorder or who have one or more cardiovascular risk factors, taking cardiovascular treatment or using doping products. The primary endpoint is the degree of correlation between course induced right ventricular functional abnormalities (by the use of 2d-strain ultrasound imaging) and the number of VEB from RV during or up to 72 hours after the race.

Procedure:

The study will take place during the Embrun triathlon in August 2019. There will be 2 evaluations: one before the race and one 30 minutes after the race, where will be carried out a self-questionnaire, a clinical examination, EKG, echocardiography and spirometry. An EKG holter in the form of a patch, adapted to sport and submersible practice, will be put in place 24 to 48 hours before the race and left until 72 hours after the race.

Outcomes / perspectives:

Characterizing the effects of a long-distance triathlon on cardiac contractile function and evaluating the athlete's rhythmic risk would make it possible to better understand these pathophysiological consequences and ultimately better detect athletes at risk of sudden death.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age between 20 to 54 years old
* Participating in the triathlon of Embrun 2019
* Collection of free and informed consent given verbally and in writing.

Exclusion Criteria:

* History of heart disease
* History of cardiac rhythm disorder.
* Subject with 1 or more cardiovascular risk factors (tobacco, diabetes, hypertension, BMI> 30).
* Cardiac, vascular or respiratory treatment(s).
* Use of substances on the list of doping products of the French Anti-Doping Agency (https://www.afld.fr/wp-content/uploads/2018/01/Liste-des- prohibitions-2018.pdf)
* Subject in relative exclusion period compared to another protocol or for which the annual amount of the maximum indemnities of 4500 € has been reached.
* Participation of the subject in another study
* Subject not affiliated to a social security scheme, or not a beneficiary of such a scheme.
* Pregnant or nursing woman, patient unable to give her protected primary consent, vulnerable persons (art.L.1121-6, L.1121-7, L.1211-8, L.1211-9)
* Subject deprived of liberty by judicial or administrative decision

Ages: 20 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Test correlation between functional of RV changes after the race and apparition of VEB | 2 or 1 day(s) before the race and 3 days after
  Test the existence of a correlation between:
  * the right ventricular functional changes observed immediately following an intense and prolonged exercise, evaluated by echocardiography and the "2d-strain" longitudinal deformation imaging technique, by performing the examination just after the race and by comparing it with before race : the main endpoint considered will be the value of the systolic peak of global longitudinal deformation (mean of the 3 segments of the free wall of the right ventricle),
  * and the number of VEB / 30 minutes from the right ventricle, quantified by an ECG holter worn during the race and up to 72 hours after the race.

SECONDARY OUTCOMES:
The secondary objectives are to characterize the respiratory impairment of this type of course and to study its relation with the functional anomalies of the RV and the occurrence of VEB. | 2 or 1 day(s) before the race and 3 days after
  Test the existence of a correlation between:
  * modification of the respiratory function (Forced expiratory volume, Carbon Monoxide gaz transfer) in comparison with after and before the race
  * and right ventricular functional changes, evaluated by echocardiography and the "2d-strain" longitudinal deformation imaging technique (value of the systolic peak of global longitudinal deformation (mean of the 3 segments of the free wall of the right ventricle) and the occurrence of VEB

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Hédon, MD, Principal Investigator — Montpellier University and Hospital
Locations (1):
- Arnaud de Villeneuve, CHU, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No